CLINICAL TRIAL: NCT07098858
Title: The WiSE®-UP Registry (The WiSE System Utilization & Performance Registry)
Status: Recruiting | Type: Observational
Sponsor: EBR Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP-10005
Record Dates: First submitted 2025-07-10; First posted 2025-08-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Single-arm, prospective, multicenter, observational study.: Market-released WiSE System approved for commercial release with a market-released co-implanted system are eligible.
  Interventions: Device: The Wise System

INTERVENTIONS:
Device: The Wise System — The WiSE CRT System is an implantable cardiac system to provide left ventricular (LV) pacing stimulation in conjunction with a co-implanted system that provides right ventricular (RV) stimulation. In combination, the devices deliver biventricular (BiV) pacing.

SUMMARY:
Observe to understand product performance, including patient safety, clinical outcomes, and CRT response information associated with the use of the market-released WiSE System

DETAILED DESCRIPTION:
The WiSE-UP Registry is a prospective, real-world, observational study aimed at understanding acute and long-term product performance, including patient safety, clinical outcomes, and CRT response information associated with the use of the market-released WiSE System.

ELIGIBILITY:
* Patient or legally authorized representative can provide written authorization and/or consent per institution requirements.
* Patient is intended to receive a WiSE System and passed the acoustic window screening
* Patient who is, or will be, accessible for follow-up.
* Participation is not excluded by local law.
* Patient is not enrolled in a concurrent drug and/or device study that may confound the Registry results.
* Patient life expectancy >1 year.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 320 patients will be enrolled in the registry and followed for five years.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2032-09-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Safety | 1, 6, 12, 24, 48 and 60 months
  The primary outcome measure of the Registry is the rate of serious adverse events (SAEs) at < 30 days post implant related to the WiSE System and/or implant procedure.

SECONDARY OUTCOMES:
Efficacy 1 | 1 month
  Procedural Success of the Leadless LV endocardial pacing (LVEP)
Efficacy 2 | 1 month
  CRT response assessment of NYHA functional classification
Efficacy 3 | 6 months
  Left ventricular ejection fraction (LVEF)
Efficacy 4 | 6 months
  Left ventricular and systolic volume (LVESV)
Efficacy 5 | 1, 6, 12, 24, 48 and 60 months
  Heart failure clinical composite score (HF CCS) categorizing patients as improved, unchanged or worsened
Efficacy 6 | 1, 6, 12, 24, 48 and 60 months
  New York Heart Association (NYHA) classification values of Markedly improved, Moderately improved, Mild improvement, No change or Slightly worse
Efficacy 7 | 1, 6, 12, 24, 48 and 60 months
  QRS duration
Efficacy 8 | 6 and 12 months
  Minnesota Living with Heart Failure Questionnaire (MLHFQ) a validated tool designed to assess the impact of heart failure on a patient's quality of life
Efficacy 9 | 1, 6, 12, 24, 48 and 60 months
  Events assessment: confirmation of reportable events including updates to any previously reported events
Efficacy 10 | 1, 6, 12, 24, 48 and 60 months
  Mortality is based on an estimated 1-year rate of 10%- and 1-year attrition of up to 15%
Efficacy 11 | 1, 6, 12, 24, 48 and 60 months
  Patient global assessment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arrhythmia Research Group (St. Bernards Hospital), Jonesboro, Arkansas
  - Naples Community Hospital, Naples, Florida